CLINICAL TRIAL: NCT02965924
Title: Effect of Topical Phenylephrine 2.5% on Episcleral Venous Pressure in Normal Human Eyes
Brief Title: Effect of Topical Phenylephrine 2.5% on EVP in Normal Human Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Arthur J. Sit, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-007077
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Assess Phenylephrine on EVP and IOP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Phenylephrine (Experimental): Subjects will receive topical phenylephrine 2.5% eye drop instilled in one eye after all baseline measurements.
  Interventions: Drug: Phenylephrine 2.5%

INTERVENTIONS:
Drug: Phenylephrine 2.5% — Instilling phenylephrine 2.5% eye drop

SUMMARY:
Phenylephrine hydrochloride ophthalmic solution is an alpha-1 adrenergic receptor agonist commonly used topically for dilation prior to ocular fundus examination. In the eye, phenylephrine acts locally as a potent vasoconstrictor and mydriatic by constricting ophthalmic blood vessels and the radial dilator muscle of the iris. Episcleral venous pressure (EVP) is a determinant of intraocular pressure (IOP) and can be measured non-invasively by venomanometry. Since phenylephrine is a vasoconstrictor, it may affect episcleral venous tone, but the effect on EVP is unknown. Understanding the physiology of episcleral veins helps us in better understanding of pathophysiology of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Any self-declared ethno-racial category.
* Medically healthy subjects.
* Subjects with two healthy eyes.
* Intraocular pressure (IOP) less than 22 mmHg in each eye.
* Best-corrected visual acuity (BCVA) in each eye 20/50 or better.
* Open angles in both eyes.
* Contact lens wear stopped at least 3 days prior to study, and during the study.
* Ability to cooperate for examinations required for study.

Exclusion Criteria:

* Chronic or acute ophthalmic diseases including glaucoma, wet type macular degeneration, uveitis and clinically significant cataract.
* Evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis.
* Cornea pathologic changes preventing reliable measurement.
* Narrow anterior chamber angle.
* Previous intraocular surgeries, laser procedures, and intravitreal injections.
* Previous corneal refractive surgeries.
* Myopia greater than -6.00 D spherical equivalent.
* Hyperopia greater than +2.00 D spherical equivalent.
* Lack of suitable episcleral vein for measurement.
* Ocular trauma within the past 6 months.
* Ocular infection or ocular inflammation in the past 3 months.
* Ocular medication of any kind within 30 days of study visit.
* Known hypersensitivity to Phenylephrine or topical anesthetic medication.
* Severe hypertension: Systolic blood pressure greater than 180 mmHg and/or diastolic blood pressure greater than 105 mmHg.
* A known history of ischemic heart disease (angina or myocardial infarction), cerebrovascular accidents, cardiac arrhythmias, cerebral or aortic aneurysms.
* Uncontrolled diabetes mellitus.
* Uncontrolled hyperthyroidism.
* Use of some systemic medications within 30 days prior to study including: β-adrenergic antagonists, α-adrenergic agonists and antagonists, calcium channel blockers, diuretics, vasodilators, monoamine oxidase inhibitors, and systemic steroids.
* Participation in any interventional study within the past 30 days prior to study visit.
* Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Sit, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenylephrine
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phenylephrine
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Episcleral Venous Pressure (EVP)
Description: EVP will be measured non-invasively using a custom-modified slit-lamp mounted venomanometer. This device utilizes the pressure chamber technique, in which a clear flexible balloon is placed against the conjunctival surface of the eye, and the pressure is increased until an episcleral vein is noted to blanch. The system for pressure-chamber based venomanometry includes a computer-controlled motor drive to increase pressure automatically, a transducer to record pressure, and a high-definition video camera to record vein collapse. Pressure measurements are synchronized with the video stream and image analysis software is used to determine the pressure required to collapse the vein to a specific pre-determined degree as measured in mmHg.
Time Frame: baseline, 60 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phenylephrine
Number analyzed (Participants) | 20
mmHg | 7.2 (2.0)
Statistical Analysis 1: Comparison: Phenylephrine; Test type: Superiority; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Change in Intraocular Pressure (IOP)
Description: Intraocular pressure will be measured in mmHg after topical anesthesia by using the pneumatonometer. There will be a minimum of three IOP measurements and a mean will be accepted as IOP.
Time Frame: baseline, 60 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phenylephrine
Number analyzed (Participants) | 20
mmHg | 15.0 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 1 year
Arm/Group | Phenylephrine
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT02965924/Prot_SAP_000.pdf